CLINICAL TRIAL: NCT05283408
Title: Effect of Dexmedetomidine and Esketamine Combined Infusion on Postoperative Pain and Recovey Quality Undergoing Modified Radical Mastectomy
Brief Title: The Clinical Study of Dexmedetomidine and Esketamine Combined Infusion Undergoing Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xuwen521
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-03

CONDITIONS: Dexmedetomidine, Esketamine, Postoperative Pain and Recovery Quality
Keywords: Dexmedetomidine; esketamine; pain; recovery quality
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine infusion on recovey quality with radical mastectomy (Experimental): Drug: Dexmedetomidine infusion Patients received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation
  Interventions: Drug: Dexmedetomidine infusion; Drug: Co-administration dexmedetomidine and low-dose esketamine infusion; Drug: Co-administration dexmedetomidine and high-dose esketamine infusion
- Co-administration dexmedetomidine and low-dose esketamine on recovey quality with radical mastectomy (Experimental): Drug: Dexmedetomidine and low-dose eskeamine combined infusion Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively.
  Interventions: Drug: Dexmedetomidine infusion; Drug: Co-administration dexmedetomidine and low-dose esketamine infusion; Drug: Co-administration dexmedetomidine and high-dose esketamine infusion
- Combined dexmedetomidine and high-dose esketamine on recovey quality with radical mastectomy (Experimental): Drug: Dexmedetomidine and high-dose eskeamine combined infusion Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively.
  Interventions: Drug: Dexmedetomidine infusion; Drug: Co-administration dexmedetomidine and low-dose esketamine infusion; Drug: Co-administration dexmedetomidine and high-dose esketamine infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Patients received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation
Drug: Co-administration dexmedetomidine and low-dose esketamine infusion — Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively.
Drug: Co-administration dexmedetomidine and high-dose esketamine infusion — Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively.

SUMMARY:
BACKGROUND: Some studies have revealed that intravenous dexmedetomidine and esketamine alleviated postoperative pain and improve the quality of recovery after surgery. The investigators investigated whether co-administration dexmedetomidine and esketamine could better alleviated postoperative pain and improve the the quality of recovery after modified radical mastectomy.

METHODS: One hundred and thirty-five women with elective modified radical mastectomy were randomly divided into 3 groups: Patients in group D received dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until 20 min before the end of operation. Patients in group DE1 received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 2 µg/kg/min until 20 min before the end of operation, respectively. Patients in group DE2 received received a bolus infusion of dexmedetomidine (0.5 µg/kg) and esketamine (0.5 mg/kg)over 10 min before the induction of anesthesia, and then dexmedetomidine were infused at a rate of 0.4 µg/kg/h and 4 µg/kg/min until 20 min before the end of operation, respectively. Primary outcome was the quality of recovery (QoR-15) at 1 day after sugery and 3 day after sugery. The secondary outcomes included perioperative remifentanil consumption, postoperative VAS pain scores, side effects such as the incidence of postoperative nausea, vomiting and bradycardia, hallucination, nightmare, as well as postoperative rescue analgesics and anti-emetics, recovery time, and extubation time.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status Ⅰ- Ⅱ
* Scheduled for elective modified radical mastectomy

Exclusion Criteria:

* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative psychiatric
* Preoperative bradycardia
* Preoperative atrioventricular block
* Preoperative hypertension
* BMI>30

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of recovery scores(QoR-15) | 1 day after operation
  Our primary outcome was quality of recovery scores(QoR-15) 1 day after operation

SECONDARY OUTCOMES:
Intraoperative remifentanil total dose | Intraoperative
  Secondary Outcome Measure was remifentanil total dose during the perioperative period
Pain visual analogue scale scores | The first 48 hours after operation
  Secondary Outcome Measure was pain visual analogue scale scores
incidence of PONV | The first 48 hours after operation
  Secondary Outcome Measure was incidence of PONV

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China